CLINICAL TRIAL: NCT00742781
Title: Vitamin D and Crohn's Disease" From the Bench to the Clinic
Brief Title: Vitamin D Supplementation in Crohn's Patients
Acronym: CTSA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Margherita T. Cantorna, Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CTSA-PPA-1
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Inflammatory Bowel Disease
Keywords: Crohn's; vitamin D
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary supplement (Experimental): Dietary supplement of vitamin D
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Oral supplementation daily with up to 5000 IU over 6 months.
  Other Names: Cholecalciferol

SUMMARY:
The purpose of this study is to determine the effect of vitamin D supplementation in Crohn's disease patients. Patients will be evaluated for increases in circulating vitamin D levels and effects on health benefits including improved bone markers, Crohn's disease activity scores, and inflammatory markers.

DETAILED DESCRIPTION:
The incidence of autoimmune diseases like inflammatory bowel disease (IBD) has increased in developed countries over the last 50 years. We propose that decreased outdoor activity and increased pollution and diets that lack adequate vitamin D have combined to create large fluctuations in vitamin D status in developed countries and especially in populations that experience winter. Experimentally we've shown that changes in vitamin D status results in more severe forms of experimental IBD. In addition, active vitamin D (1,25(OH)2D3) completely blocks the development of experimental IBD. The vitamin D hypothesis proposes that vitamin D regulates the development and function of the immune system and that changes in vitamin D status affect the development of the resultant immune response and the development of diseases like IBD. Our hypothesis is that because of low dietary vitamin D intakes and malabsorption of many nutrients, Crohn's patients will have low circulating vitamin D levels that are detrimental for their health. We plan to give Crohn's patients 1000 IU of vitamin D/d and determine whether this dose is well tolerated, induces an increase in circulating vitamin D levels and has any additional health benefits (improved bone markers, Crohn's disease activity scores, inflammatory markers).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years of age with mild to moderate Crohn's disease who are not on active steroid treatment and who do not have ostomies.

Exclusion Criteria:

* Patients with ulcerative colitis or other bowel conditions which are not Crohn's.
* Patients with ostomies.
* Those currently using supplemental vitamin D in excess of the amount in one multivitamin per day.
* Regular tanning bed users.
* Persons who report more than moderate alcohol consumption ( > 1 drink/day for women > 2 for men).
* Pregnant or lactating women or women planning a pregnancy during the study time frame.
* Regular users of medications which may interfere with assessment of study outcomes .
* Those who cannot understand written or spoken English .
* Individuals under medical psychiatric care.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-05; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margherita T Cantorna, PhD, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Pennsylvania State University, University Park, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited form the Pennsylvania State University University Park area and Hershey College of Medicine. The University General Clinical Research Centers on the two campuses were utilized. Recruitment was from 5/2009 to 7/2011.
Pre-assignment Details: The study was an open label feasibility study that used patients as their own controls. All patients were accepted into the study as long as they met the eligibility requirements.
Period: Overall Study
Arm/Group | Vitamin D Supplementation
Started | 21
Completed | 18
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D Supplementation
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Crohn's Disease Activity Index
Description: Questionnaire and physical measurements combine to generate a score. Scores below 150 indicate remission, 150-350 mild to moderate disease, over 350 severe disease. The total range of scores are from 0- Don't have Crohn's disease to 600 severe Crohn's disease. 0-150 is remission, 151-219 is mild, 220-450 is moderate disease and over 451 is severe.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Vitamin D Supplemented
Number analyzed (Participants) | 21 | 18
units on a scale | 230 (74) | 112 (81)

2. Secondary Outcome: Health Improvement
Description: International Physical Activity Questionnaire. Minutes/week for 30 min/day, 5days (MET) are calculated for different activity intensities. Total range of scores 0-600 MET low activity, 600-1200 Moderate activity, Over 1200-3000 High activity.
Time Frame: 6 months
Population: Activity records for 14 participants were recorded at baseline and after vitamin D supplementation.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Vitamin D Supplemented
Number analyzed (Participants) | 14 | 14
units on a scale | 5778 (969) | 6714 (1327)

3. Primary Outcome: 25(OH)D3 Serum Levels
Description: 25(OH)D3 levels before and after vitamin D supplementation.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ng/ml 25(OH)D3
Arm/Group | Baseline | Vitamin D Supplemented
Number analyzed (Participants) | 21 | 18
ng/ml 25(OH)D3 | 16 (10) | 45 (19)

ADVERSE EVENTS:
Time Frame: The period when adverse outcomes for each individual was 7 months.
Description: No adverse events were noted in any of the patients.
Arm/Group | Vitamin D Supplemented
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
The main limitation of the study was the lack of placebo control and the small size of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No